CLINICAL TRIAL: NCT00186108
Title: A Pilot Study Evaluating Oral Triamcinalone in Patients With Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROS0006
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Prostate Cancer
Keywords: Oral Triamcinalone; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oral Triamcinalone

SUMMARY:
The primary purpose of this study is to evaluate the ability of oral triamcinalone given twice a day to patients with androgen independent prostate cancer to produce a sustained biochemical response. Secondary goals are to describe the safety and tolerability at this dose and schedule, to determine the time to sustained biochemical response, to determine the duration of biochemical response, to determine the time to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Histologically documented adenocarcinoma of prostate
* Currently receiving LHRH agonists with castrate levels of testosterone or who have had an orchiectomy
* Must have had a rise in PSA despite anti androgen withdrawal
* Exhibit 2 consecutive rise in PSA after the last hormonal manipulation
* Minimum PSA of greater than 5 KPS greater than 80%
* Normal cortisol level at entry
* Life expectancy greater than 6 months
* Provide written consent pursuant to regulatory requirements prior to initiation of study procedure

Exclusion criteria:

* Younger than 18 years
* Patients without prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Ability of oral triamcinalone given twice a day to patients with androgen independent prostate cancer to produce a sustained biochemical response. | Following treatment

SECONDARY OUTCOMES:
Safety and tolerability at this dose and schedule, time to sustained biochemical response, duration of biochemical response, time to disease progression | Following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Srinivas, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Center, Stanford, California, United States